CLINICAL TRIAL: NCT04442191
Title: Infusion of Convalescent Plasma for the Treatment of Patients Infected With Severe Acute Respiratory Syndrome-Coronavirus-2 (COVID-19): A Double-blinded, Placebo-controlled, Proof-of-concept Study
Brief Title: Convalescent Plasma as a Possible Treatment for COVID-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jesica Herrick, Assistant Professor of Clinical Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0441
Record Dates: First submitted 2020-05-11; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient's nurse will be instructed to place the blood product in a paper bag so the label on the product is not visible to the study physicians or to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): This study will utilize convalescent plasma from donors recovered from infection with SARS-CoV-2 (which causes COVID-19) with neutralizing antibody titers >1:64.
  Interventions: Biological: Convalescent plasma
- Placebo (Placebo Comparator): Placebo utilized in this study will include Fresh Frozen Plasma collected before the COVID-19 pandemic began. As an extra control, some of this plasma will be saved and tested for COVID-19 antibodies to ensure they are not present.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Convalescent plasma — This study will use convalescent plasma collected from those who have previously had COVID-19 and have been shown to have cleared the infection and made antibodies against the virus.
  Other Names: Fresh Frozen Plasma
  Arms: Convalescent plasma
Biological: Placebo — The placebo arm of this study will use fresh frozen plasma that presumably does not contain antibodies against COVID-19.
  Other Names: Fresh Frozen Plasma
  Arms: Placebo

SUMMARY:
Patients who are ill with COVID-19 may benefit from receiving convalescent plasma infusions containing antibodies from donors who have recovered from the disease and are proven to no longer be infected. Given the current public health emergency due to COVID-19, the FDA has recently fast-tracked the use of convalescent plasma. The purpose for this study is to assess if convalescent plasma collected from donors previously infected with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), the virus that causes COVID-19, can provide clinical benefit to those acutely ill with the virus and to evaluate if such treatment is safe.

There will be two arms in the interventional study, where subjects will either be treated with convalescent plasma or fresh frozen plasma in a randomized and blinded manner. As an additional comparison, the clinical course of subjects enrolled during the period of the study who do not receive an alternative treatment for COVID-19 will be assessed.

DETAILED DESCRIPTION:
Study Design and Procedures - Comparison group (no-treatment control)

1. Subjects will be identified by reviewing a REDCap database containing the list of all patients at the University of Illinois at Chicago Hospital (UIC) who were tested for COVID-19. Using these data, the investigators will identify those subjects who are >40 years old, were admitted to the hospital during the period of the study, otherwise met all of the inclusion and exclusion criteria for the infusion arm of the study but were not enrolled and did not receive any medications for treatment of COVID-19 (were treated with only supportive care).
2. Clinical data from the hospital admissions of these subjects will be entered into a REDCap database. The same clinical information captured for subjects who underwent transfusion (vital signs, oxygen status, etc.) will be entered into this database.

Study Design and Procedures - Intervention arms Screening Visit

1. Patients admitted to UIC Hospital and meeting the inclusion criteria will be enrolled after documentation of informed consent.
2. Enrolled subjects will answer a symptom screen, undergo a physical exam, and have clinical data extracted from their chart (including medical history, demographic information, vital signs and documentation of oxygen requirement).
3. Women of childbearing age will be asked if there is a chance that they might be pregnant, if they are currently breastfeeding, and if they are planning to become pregnant.
4. Blood will be drawn for a Complete Blood Count (CBC) and blood type and screen, and a sample of blood will be stored for research purposes.
5. Nasopharyngeal and/or oropharyngeal swabs will be collected for Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) testing.
6. A study investigator will ask the patient's primary team if they are planning on treating the patient with Remdesivir. If the patient qualifies for this medication, the study investigator will monitor the patient's chart and work with the patient's nurse to ensure that the first convalescent plasma infusion and first dose of Remdesivir are given within 24 hours of each other.

Study Design and Procedures - Transfusion Visits (Study days 0 and 1) Note - the first transfusion visit may be done on the same day as the screening visit if time permits, otherwise it will be done the following day. Items 1 and 2 will only be performed for the first transfusion visit if the visit occurs the day after the screening visit.

1. The patient's clinical status, oxygen requirement, vital signs, and physical exam will be extracted from their clinical chart. Extracted information will include:

   1. imaging: chest X-ray or chest CT results
   2. labs: CBC with differential, C-Reactive Protein (CRP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, creatinine.
   3. Demographic and medical information: history of present infection (length of symptoms prior to presentation, etc.)
2. Participants will be asked a symptom questionnaire.
3. Randomization to convalescent plasma or fresh frozen plasma will be 1:1. Randomization will be conducted by a physician not involved in the study and using pre-prepared lists with random permuted blocks of varying sizes. This physician will hand-deliver an order sheet for either convalescent or fresh frozen plasma to the blood bank (this way no orders that could potentially unblind study personnel will be in participants' charts).
4. The blood bank technical staff will select either two compatible blood-type non-therapeutic units of plasma or two compatible units of convalescent plasma, depending on which group the patient has been randomized to.
5. If the blood bank does not have any product of that patient's blood type, investigators will not be able to have the subject complete the remainder of the study. However, the investigators will keep the information about the participant's blood type in the study database. Then, in the event that plasma of the appropriate blood type is obtained, study investigators may contact participants to find out if they are still interested in being part of the study.
6. The blood product will be delivered to the floor and the participant's nurse will infuse and document plasma administration following UIC Hospital policy "TX 5.03." Study subjects will receive 1 unit of plasma the first day, with the second unit being given the next day.
7. Once the blood product has been hung, the patient's nurse will place it in a bag that will prevent the patient or physician's taking care of the patient from seeing whether the unit is regular frozen plasma or convalescent plasma. The nurse will be under instructions not to convey information about which type of plasma was used to the study team.
8. The nurse will be instructed to stop the transfusion while a small sample of plasma remains in the bag. The bag will then be sent back to the blood bank (this is usual protocol for blood products), and remaining plasma will be emptied into a storage container, labeled with the patient's study identification number, and frozen for later use for research purposes.
9. If a transfusion reaction occurs the transfusion will be stopped and reported to the blood bank as stated in UIC Hospital policy "TX 5.03."

Study Design and Procedures - Post-infusion monitoring

1. Post-transfusion clinical data will be collected from electronic medical record daily for days 2-8 following the first transfusion (or until the participant is discharged if they are discharged prior to 8 days following transfusion). This information includes:

   1. vital signs: temperature, blood pressure, respiratory rate, pulse
   2. symptoms: cough, dyspnea, shortness of breath
   3. oxygenation: oxygen saturation, supplemental oxygen requirement, supplemental oxygen method (e.g., ventilator, nasal canula, prone positioning, etc.)
   4. imaging: chest X-ray or chest CT results
   5. labs: CBC with differential, CRP, ALT, AST, total bilirubin, creatinine (and whether or not the patient has required renal support)
   6. medications: antibiotics and anti-viral medications, neuromuscular blocking agents, vasopressors
   7. location: intensive care unit, discharged, regular hospital bed
2. The participant will have a swab sample for SARS-CoV-2 RT-PCR collected daily for days 2-8 following the first transfusion (or as many days as they are admitted if they are discharged prior to 8 days following the first transfusion) and on day 14 following plasma infusion.

   Participants will also have blood drawn on days 2, 4, and 8 following the first plasma infusion for measurement of antibody titers to SARS-CoV-2 (if they are discharged prior to day 4 or 8 they will not undergo that day's blood draw).
3. If the patient is discharged prior to 14-days following infusion of plasma, they will be asked to return to Project Wish on day 14 post- infusion of plasma for a blood draw (for antibody titers), a nasopharyngeal and/or oropharyngeal swab (for RT-PCR testing) and to answer a short symptom questionnaire.
4. The patient will be contacted by telephone (if discharged) at 28-days following plasma infusion and will be asked a symptom questionnaire. If they remain in the hospital at this time point, they will be asked this questionnaire (if capable) and will have information regarding their clinical condition extracted from their chart.

ELIGIBILITY:
Inclusion Criteria:

* Patients 40 years-old and over who are admitted to the University of Illinois Hospital (UIC) due to COVID-19
* Positive oropharyngeal and/or nasopharyngeal swab test for SARS-CoV-2 by RT-PCR within the preceding 72 hours (performed by University of Illinois Hospital Laboratories or, if performed elsewhere, documented in the patient's UIC medical record)
* Symptomatic infection with any of the following: fever, cough, dyspnea, or tachypnea > 22 breaths/min
* Need for supplemental oxygen, between 1-5 liters/minute by nasal canula, to maintain O2 saturations >92%
* Consents to comply with all protocol requirements
* Agrees to storage of specimens for future testing

Exclusion Criteria:

* Patients with known Immunoglobulin A deficiency (high risk of severe or fatal anaphylactic reactions)
* Patients who are on a ventilator
* Patients with past history of severe transfusion reaction including transfusion-related acute lung injury (TRALI) or anaphylaxis
* Patients with a baseline requirement for supplemental oxygen due to chronic lung disease or with known history of either moderate-to-severe asthma or emphysema.
* Female subjects who report that they are pregnant or breastfeeding
* Receipt of pooled immunoglobulin in the past 30 days
* Patients must be willing to not take any another alternative experimental treatment for COVID-19 from the time they undergo enrollment until the 28-day follow-up phone call

  •. Participants who are being treated with Remdesivir and have had their first dose of Remdesivir greater than 24 hours prior to the time they will receive their first dose of convalescent plasma
* Patients with severe disease due to COVID-19, as manifested by a need for vasopressors, and/or diagnosis of Acute Respiratory Distress Syndrome

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-05-05 (Estimated)

PRIMARY OUTCOMES:
Oxygen supplementation | 8 days
  The primary endpoint will be clinical response at 8 days, defined as no need for oxygen supplementation for the previous 24 hours.

SECONDARY OUTCOMES:
28-day and in-hospital mortality rate | 28 days
  Mortality rate during the 28 days of follow-up and during the subjects' initial hospital stays
Number of participants transferred to the Intensive Care Unit (ICU) | 28 days
  Transfer to an ICU bed during the 28 days following study enrollment
Number of participants intubated | 28 days
  Intubation within the 28 days following study enrollment
Length of hospital stay in days | 28 days
  Number of days admitted to the hospital during the 28-day follow-up period
Type of respiratory support | 28 days
  Type of respiratory support required during the 28-day follow-up period: intubation, high-flow oxygen by nasal canula, nasal canula
C-reactive Protein (CRP) | 28 days
  Change in CRP following treatment
Lymphocyte count | 28 days
  Change in lymphocyte count following treatment
Length or respiratory support required, in days | 28 days
  Number of days respiratory support is required
Lactate dehydrogenase (LDH) | 28 days
  Change in LDH following treatment
Ferritin | 28 days
  Change in Ferritin level following treatment
D-Dimer | 28 days
  Change in D-Dimer level following treatment
White Blood Cell (WBC) Count | 28 days
  Change in WBC count following treatment

OTHER OUTCOMES:
Safety endpoint: Severe transfusion reaction | 6 hours following transfusion
  Severe transfusion reaction will be defined as having any of the following occur within 6 hours of the infusion of blood product and not attributable to the underlying disease: 1) an increase of 2 L/minutes or more in supplemental oxygen requirement compared to the baseline requirement before transfusion, 2) oxygen saturations <93% despite oxygen via nasal canula, or 3) need for transfer to the ICU.
Safety endpoint two: adverse events | 24 hours following transfusion
  Cumulative incidence of adverse events during the study period: transfusion reaction (fever, rash), transfusion related acute lung injury (TRALI), transfusion associated circulatory overload (TACO), transfusion related infection.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No